CLINICAL TRIAL: NCT02551666
Title: Balance Recovery Training for Fall Prevention in Retirement Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other); University of Michigan (Other)
Responsible Party: Principal Investigator, Michael Madigan, Professor, Biomedical Engineering, Texas A&M University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TexasAMU
Record Dates: First submitted 2015-08-12; First posted 2015-09-16 (Estimated); Results first posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-06

CONDITIONS: Accidental Falls, Aged, Exercise Movement Techniques
MeSH Terms: interventions — Aquatic Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Tai Chi exercise intervention (Active Comparator): Participants will perform 30-minute Tai Chi sessions (Yang Short form) 3 times a week for 4 weeks.
  Interventions: Other: Tai Chi exercise
- Balance recovery training (Experimental): Participants will practice balance recovery on a modified treadmill for approximately 30-minutes per session, 3 sessions a week for 4 weeks.
  Interventions: Other: Balance recovery training

INTERVENTIONS:
Other: Balance recovery training — Participants will practice recovering their balance after a perturbation similar to tripping while walking. Each of these 'balance recovery training' sessions will last approximately 30 minutes, and will be performed 3 times per week for 4 weeks.
  Arms: Balance recovery training
Other: Tai Chi exercise — Participants will perform Tai Chi exercises (Yang short form) for 30 minutes, 3 times a week for 4 weeks. Each session will be led by an experienced Tai Chi instructor.
  Arms: Tai Chi exercise intervention

SUMMARY:
Falls are the leading cause of injuries and injury-related deaths among older adults over the age of 65 in the United States. To help reduce the number of these falls, there is growing interest in using reactive balance training to improve the reactive response to common perturbations (e.g., tripping and slipping). The goal of this study was to compare treadmill-based reactive balance training versus Tai Chi performed at, and among residents of, older adult senior housing. We hypothesized that participants randomized to reactive balance training (RBT) would show better performance on reactive balance tests compared to participants randomized to Tai Chi. We also hypothesized that participants randomized to Tai Chi would show better performance on clinical tests of balance and mobility compared to participants randomized to RBT. The long-term goal of this work is to demonstrate the value of RBT over Tai Chi for preventing falls resulting from sudden, external perturbations.

Thirty-five residents of five senior housing facilities were allocated to either treadmill-based reactive balance training or Tai Chi training. Both interventions were performed three times per week for four weeks, with each session lasting approximately 30 minutes. A battery of balance tests was performed at baseline, and again one week, one month, three months, and six months post-training. The battery included six standard clinical tests of balance and mobility, and a test of reactive balance performance.

ELIGIBILITY:
Inclusion Criteria:

* Must be age 70 or older
* Must be a resident of local continuing care retirement community (CCRC)
* Must be able to walk down a long hallway without any aids (cane, walker, etc.)
* Must not have a fragility fracture in the past 10 years
* Must not smoke
* Must not be in physical therapy
* Must not perform more than 150 minutes/week of moderate to vigorous aerobic activity
* Must score 24 or higher on Folstein Mini Mental Status Exam
* Must have less than 20% probability of major osteoporotic fracture as assessed by the fracture risk assessment tool (FRAX) score
* Must not have recently (within 1 year) participated in Tai Chi

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Madigan, PhD, Principal Investigator — Virginia Polytechnic Institute and State University

IPD SHARING:
Plan to Share IPD: Yes
All outcome measures at the time points described above will be shared with other researchers.
Supporting Information: Study Protocol, ICF
Time Frame: These data will be made available starting one year after publication.
Access Criteria: Access will be provided for supplementary analyses. IPD will be shared via email.

REFERENCES:
- [Result] Madigan ML, Aviles J, Allin LJ, Nussbaum MA, Alexander NB. A Reactive Balance Rating Method That Correlates With Kinematics After Trip-like Perturbations on a Treadmill and Fall Risk Among Residents of Older Adult Congregate Housing. J Gerontol A Biol Sci Med Sci. 2018 Aug 10;73(9):1222-1228. doi: 10.1093/gerona/gly077. PMID 29668910

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 151 prospective subjects were assessed for eligibility. 74 failed the medical screening 28 ended up declining to participate after learning more about the study 14 were withdrawn for other reasons not related to the study
  35 participants remained and were allocated to one of the two treatment groups.
Groups:
- Tai Chi Exercise: Participants performed 30-minute Tai Chi sessions (Yang Short form) 3 times a week for 4 weeks.
  Tai Chi exercise: Participants performed Tai Chi exercises (Yang short form) for 30 minutes, 3 times a week for 4 weeks. Each session was be led by an experienced Tai Chi instructor.
- Balance Recovery Training: Participants performed balance recovery on a modified treadmill for approximately 30-minutes per session, 3 sessions a week for 4 weeks.
  Balance recovery training: Participants practiced recovering their balance after a perturbation similar to tripping while walking. Each of these 'balance recovery training' sessions lasted approximately 30 minutes, and was performed 3 times per week for 4 weeks.
Period: Overall Study
Arm/Group | Tai Chi Exercise | Balance Recovery Training
Started | 16 | 19
Completed | 15 | 16
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tai Chi Exercise Intervention | Balance Recovery Training | Total
Number analyzed (Participants) | 16 | 19 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 82.6 (4.5) | 80.9 (6.2) | 81.7 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 5 | 6 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 16 | 19 | 35
Body mass index (kg/m^2) [Mean (Standard Deviation); unit: kg/(m^2)] | 30.8 (4.5) | 28.6 (5.3) | 29.6 (5.0)
Number of participants reporting falls with injury in the past year [Number; unit: participants] | 5 | 1 | 6
Number of participants reporting 2 or more falls in the past year [Number; unit: participants] | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Maximum Torso Angle at 0.8 Mph
Description: maximum torso angle during a simulated trip, and be measures in degrees. Larger angles indicate worse performance.
Time Frame: 1 week, 1 month, 3 months, and 6 months after completing four weeks of exercise intervention
Population: participants who completed at least 9 of 12 sessions
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Tai Chi Exercise | Balance Recovery Training
Number analyzed (Participants) | 16 | 19
degrees
  Baseline | 18.8 (9.0) | 23.9 (10.6)
  1 week post intervention | 20.5 (8.8) | 11.7 (4.4)
  1 month post intervention | 17.5 (7.1) | 13.1 (5.7)
  3 months post intervention | 16.8 (3.6) | 13.0 (4.1)
  6 months post intervention | 18.2 (7.5) | 16.2 (10.5)

2. Primary Outcome: Maximum Torso Angle at 1.6 Mph
Description: maximum torso angle during a simulated trip, and be measures in degrees. Larger angles indicate worse performance.
Time Frame: 1 week, 1 month, 3 months, and 6 months after completing four weeks of exercise intervention
Population: participants who completed at least 9 of 12 sessions
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Tai Chi Exercise | Balance Recovery Training
Number analyzed (Participants) | 16 | 19
degrees
  Baseline | 29.7 (14.1) | 28.4 (10.4)
  1 week post intervention | 29.6 (12.0) | 21.7 (10.8)
  1 month post intervention | 22.2 (6.2) | 23.0 (12.3)
  3 months post intervention | 28.8 (7.8) | 26.9 (16.5)
  6 months post intervention | 27.1 (12.5) | 24.2 (9.8)

3. Secondary Outcome: Reactive Balance Rating
Description: The reactive balance rating evaluates performance in response to six separate tests on a treadmill involving sudden acceleration of the belt to elicit a loss of balance from stance. The administrator scores as 0, 1, or 2: a) the overall effectiveness of the initial stepping response to each treadmill acceleration, and b) the amount of support provided by the harness or spotter next to the participant. These scores are then combined using a rubric to determine the overall reactive balance rating.
  The reactive balance rating is a score on a scale from 0 to 12 where higher scores indicates a better outcome.
  More details are available at: Madigan ML, Aviles J, Allin LJ, Nussbaum MA, Alexander NB. A Reactive Balance Rating Method That Correlates With Kinematics After Trip-like Perturbations on a Treadmill and Fall Risk Among Residents of Older Adult Congregate Housing. The Journals of Gerontology: Series A. 2018: 73(9): 1222-1228.
Time Frame: 1 week, 1 month, 3 months, and 6 months after completing four weeks of exercise intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tai Chi Exercise | Balance Recovery Training
Number analyzed (Participants) | 16 | 19
score on a scale
  Baseline | 4.3 (2.0) | 4.8 (3.5)
  1 week after intervention | 6.3 (2.4) | 8.2 (3.2)
  1 month after intervention | 6.1 (3.3) | 8.7 (3.2)
  3 months after intervention | 7.1 (2.4) | 8.0 (3.2)
  6 months after intervention | 6.7 (2.2) | 8.1 (3.6)

4. Secondary Outcome: Step Length at 0.8 Mph
Description: step length during reactive balance trial.
Time Frame: 1 week, 1 month, 3 months, and 6 months after completing four weeks of exercise intervention
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Tai Chi Exercise | Balance Recovery Training
Number analyzed (Participants) | 16 | 19
meters
  Baseline | .49 (.06) | .51 (.09)
  1 week post intervention | .44 (.12) | .52 (.09)
  1 month post intervention | .48 (.09) | .51 (.08)
  3 months post intervention | .50 (.08) | .52 (.12)
  6 months post intervention | .49 (.11) | .53 (.07)

5. Secondary Outcome: Timed-up-and-go Test
Description: The timed-up-and-go tests is measured in seconds. Longer times indicate worse performance.
Time Frame: 1 week, 1 month, 3 months, and 6 months after completing four weeks of exercise intervention
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Tai Chi Exercise | Balance Recovery Training
Number analyzed (Participants) | 16 | 19
seconds
  Baseline | 14.8 (6.0) | 12.9 (4.5)
  1 week post intervention | 13.6 (3.9) | 12.1 (3.7)
  1 month post intervention | 13.2 (4.2) | 11.8 (3.6)
  3 months post intervention | 11.9 (3.4) | 11.7 (3.7)
  6 months post intervention | 13.2 (4.7) | 12.2 (4.3)

6. Secondary Outcome: Unipedal Stance Time Test
Description: The unipedal stance time is measured in seconds, up to a maximum of 30 seconds. Longer times indicate better performance.
Time Frame: 1 week, 1 month, 3 months, and 6 months after completing four weeks of exercise intervention
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Tai Chi Exercise | Balance Recovery Training
Number analyzed (Participants) | 16 | 19
seconds
  Baseline | 4.0 (3.2) | 5.7 (6.4)
  1 week post intervention | 6.0 (4.9) | 6.3 (7.4)
  1 month post intervention | 5.3 (4.5) | 7.6 (10.4)
  3 months post intervention | 4.8 (3.7) | 6.8 (9.8)
  6 month post intervention | 8.3 (8.7) | 6.5 (9.7)

7. Secondary Outcome: Maximum Step Length Test
Description: Maximum step length is measured in inches. Longer maximum step length indicates better performance.
Time Frame: 1 week, 1 month, 3 months, and 6 months after completing four weeks of exercise intervention
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Tai Chi Exercise | Balance Recovery Training
Number analyzed (Participants) | 16 | 19
inches
  Baseline | 18.1 (5.2) | 20.5 (5.7)
  1-week post intervention | 18.9 (3.6) | 21.0 (3.2)
  1-month post intervention | 18.9 (5.7) | 22.5 (3.7)
  3-month post intervention | 20.7 (4.3) | 20.4 (3.2)
  6-month post intervention | 20.8 (5.0) | 20.7 (3.6)

8. Secondary Outcome: Activities-specific Balance Confidence (ABC) Scale
Description: Activities-specific balance confidence scale ranges from 0 to 100. Larger values indicate more confidence (i.e. better outcome).
Time Frame: 1 week, 1 month, 3 months, and 6 months after completing four weeks of exercise intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tai Chi Exercise | Balance Recovery Training
Number analyzed (Participants) | 16 | 19
score on a scale
  Baseline | 76.2 (16.3) | 74.0 (14.1)
  1-week post intervention | 79.3 (15.4) | 76.6 (13.8)
  1-month post intervention | 78.1 (13.8) | 78.9 (12.0)
  3-months post intervention | 76.9 (13.9) | 75.7 (12.9)
  6-months post intervention | 76.0 (17.9) | 76.6 (12.0)

9. Secondary Outcome: Performance-oriented Mobility Assessment (POMA)
Description: The Performance-oriented Mobility Assessment is a common clinical test for assessing a person's static and dynamic balance abilities. The test is in two short sections that contain one examining static balance, and the other gait. The section examining static balance includes 9 individual tests scored 0, 1, or 2 by the test administrator based upon their observation of the balance performance (higher is better). The section on gait includes 7 individual tests scored 0, 1, or 2 by the test administrator based upon their observation of the gait performance (higher is better). All of these individual test scores are then summed to determine the overall Performance-oriented Mobility Assessment score.
  The overall Performance-oriented Mobility Assessment score is on a scale from 0 to 28. Larger values indicate better mobility.
  Additional details are published here: Tinetti ME. Performance-oriented assessment of mobility problems in elderly patients. JAGS 1986; 34: 119-126.
Time Frame: 1 week, 1 month, 3 months, and 6 months after completing four weeks of exercise intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tai Chi Exercise | Balance Recovery Training
Number analyzed (Participants) | 16 | 19
score on a scale
  Baseline | 23.4 (2.9) | 23.7 (2.8)
  1-week post intervention | 24.9 (2.4) | 23.9 (2.0)
  1-month post intervention | 24.1 (2.8) | 24.9 (1.7)
  3-month post intervention | 24.5 (2.3) | 24.9 (2.6)
  6-month post intervention | 23.1 (3.3) | 24.3 (2.4)

10. Secondary Outcome: Berg Balance Test
Description: The Berg balance test is measures that evaluates static balance and fall risk using 14 individual sub-tests. It includes static and dynamic activities of varying complexity. The test administrator scores performance on each sub-test as either a 0, 1, 2, 3, or 4. All scores are sub-tests are then summed to determine the overall Berg balance test score.
  The Berg balance test score is on a scale from 0 to 56. Larger values indicate better balance.
  More information is available at: Berg, K., Wood-Dauphine, S.L. and Williams, J.L. Measuring balance in the elderly: validation of an instrument. Can. J. Public Health, 83(S2): S7-S11, 1992.
Time Frame: 1 week, 1 month, 3 months, and 6 months after completing four weeks of exercise intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tai Chi Exercise | Balance Recovery Training
Number analyzed (Participants) | 16 | 19
score on a scale
  Baseline | 44.5 (5.6) | 47.3 (4.3)
  1-week post intervention | 48.0 (4.5) | 48.2 (3.7)
  1-month post intervention | 47.7 (5.3) | 49.7 (3.0)
  3-month post intervention | 48.7 (4.5) | 49.0 (3.8)
  6-month post intervention | 47.7 (5.6) | 49.1 (4.5)

11. Secondary Outcome: Step Length at 1.6 Mph
Description: step length during reactive balance trial.
Time Frame: 1 week, 1 month, 3 months, and 6 months after completing four weeks of exercise intervention
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Tai Chi Exercise | Balance Recovery Training
Number analyzed (Participants) | 16 | 19
meters
  Baseline | .61 (.10) | .56 (.11)
  1 week post intervention | .56 (.10) | .62 (.09)
  1 month post intervention | .58 (.06) | .60 (.09)
  3 months post intervention | .64 (.03) | .62 (.07)
  6 months post intervention | .63 (.05) | .61 (.09)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from each participant for 28 weeks. This time period spanned from the initial baseline balance assessment to six months after completing the assigned intervention.
Description: Definition does not differ.
Arm/Group | Tai Chi Exercise | Balance Recovery Training
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/19
Other Adverse Events (participants affected / at risk) | 0/16 | 0/19

LIMITATIONS AND CAVEATS:
Sample size was not sufficient to investigate falls as an outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Informed Consent Form (2015-10-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT02551666/ICF_000.pdf
  • Statistical Analysis Plan (2015-10-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT02551666/SAP_001.pdf
  • Study Protocol (2015-10-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT02551666/Prot_002.pdf